CLINICAL TRIAL: NCT02405520
Title: A Phase I Randomized, Double-Blinded, Placebo Controlled Study to Evaluate the Safety and Immunogenicity of the Recombinant (E.Coli) Human Papillomavirus Type 6/11 Bivalent Vaccine in Healthy Volunteers Aged 18-55 Years
Brief Title: Safety and Immunogenicity Study of the Recombinant Human Papillomavirus Virus Type 6/11 Bivalent Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Xiamen University
Organization: Xiamen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPV-PRO-004
Record Dates: First submitted 2015-03-25; First posted 2015-04-01 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Condylomata Acuminata
Keywords: human papillomavirus vaccine; condylomata acuminata
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- low dosage HPV Vaccine (Experimental): Participants in this arm would receive low dosage of HPV vaccines.
  Interventions: Biological: low dosage HPV Vaccine
- medium dosage HPV Vaccine (Experimental): Participants in this arm would receive medium dosage of HPV vaccines.
  Interventions: Biological: medium dosage HPV Vaccine
- high dosage HPV Vaccine (Experimental): Participants in this arm would receive high dosage of HPV vaccines.
  Interventions: Biological: high dosage HPV Vaccine
- Placebo (Placebo Comparator): Participants in this arm would receive placebo (Aluminium Adjuvant).
  Interventions: Biological: Aluminium Adjuvant

INTERVENTIONS:
Biological: low dosage HPV Vaccine — Participants would intramuscularly receive low dosage of HPV 6/11 bivalent vaccine at 0, 1, 6 month for 3 doses.
  Arms: low dosage HPV Vaccine
Biological: medium dosage HPV Vaccine — Participants would intramuscularly receive medium dosage of HPV 6/11 bivalent vaccine at 0, 1, 6 month for 3 doses.
  Arms: medium dosage HPV Vaccine
Biological: high dosage HPV Vaccine — Participants would intramuscularly receive high dosage of HPV 6/11 bivalent vaccine at 0, 1, 6 month for 3 doses.
  Arms: high dosage HPV Vaccine
Biological: Aluminium Adjuvant — Participants would intramuscularly receive aluminium adjuvant at 0, 1, 6 month for 3 doses.
  Arms: Placebo

SUMMARY:
This phase I clinical study was designed to evaluate the safety and immunogenicity of the novel recombinant HPV type 6/11 bivalent vaccine, manufactured by Xiamen Innovax Biotech CO., LTD., in healthy volunteers aged over 18-55 years of age at enrollment. The study volunteers will receive the 3 different formulations of the novel HPV vaccine or placebo administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion criteria:

1. Health people aged between 18 and 55 years.
2. Judged as healthy and eligible for vaccination by the investigators through a self-reported medical history and some physical examinations.
3. Written informed consent was obtained from the participants.
4. Able to comply with the requests of the study.
5. Axillary temperature not higher than 37.0°C
6. Men, or non-pregnant women verified by a urine pregnancy test.

Exclusion criteria:

1. Pregnant or breastfeeding or plan to be pregnant within 7 months.
2. Use of any investigational product or non-registered product (drug or vaccine) within 30 days preceding the first dose of the study vaccine or plan to use during the study period.
3. Received immunosuppressed, immunoregulation therapy, or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment.
4. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine or plan to use within 7 months.
5. Administration of any attenuated live vaccines within 21 days preceding the first dose of the study vaccine or any subunit or inactivated vaccines within 14 days before vaccination.
6. Had a fever (axillary temperature over 38°C) within 3 days or acute illness requiring systemic antibiotics or antiviral treatment within 5 days before vaccination.
7. Having the plan to participate another clinical trial during the study period.
8. Received another HPV vaccine.
9. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, .or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response).
10. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy, urticaria, dyspnea, angioneurotic edema or abdominal pain.
11. Asthma that required emergent treatment, hospitalization, oral or intravenous corticosteroid for unstable condition within the past 2 years.
12. Having serious disease of internal medicine, such as hypertension, cardiac disease, diabetes, hyperthyroidism et al.
13. Diagnosed coagulant function abnormality (i.e., clotting factors absent, clotting hemorrhagic disease, abnormal platelet function) or blood coagulation disorder.
14. Epilepsy, except fever epilepsy at under 2 years of age, alcohol-induced epilepsy in 3 years before abstinence, or idiopathic epilepsy requiring no treatment in the past 3 years.
15. Past or current two-stage affective psychosis, not well controlled in the past 2 years or requiring drugs, or h a tendency to commit suicide.
16. Other medical, psychological, social or occupational factors that, according to the investigators' judgment, might affect the individual's ability to obey the protocol or sign the informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Measure adverse reactions/events throughout the study | 10 month
  With composite measure: Measure solicited local/systematic adverse reactions within 7 days after each vaccination; Measure unsolicited adverse reactions within 30 days after vaccination; Measure blood, liver and kidney function changes pre- and 2 days post vaccination; Measure serious adverse events occurred throughout the study

SECONDARY OUTCOMES:
Measure anti-HPV 6/11 antibody in serum samples at 7 month to evaluate the immunogenicity of the HPV 6/11 vaccine formulations. | 7 month

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Master, Study Chair — Xiamen University; Zhao-Jun Mo, Master, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control; Ting Wu, Ph. D, Study Director — Xiamen University

REFERENCES:
- [Derived] Mo ZJ, Bi ZF, Sheng W, Chen Q, Huang T, Li MQ, Cui XL, Wangjiang YH, Lin BZ, Zheng FZ, Sun G, Li YF, Zheng Y, Zhuang SJ, Su YY, Pan HR, Huang SJ, Wu T, Zhang J, Xia NS. Safety and immunogenicity of an Escherichia coli-produced bivalent human papillomavirus type 6/11 vaccine: A dose-escalation, randomized, double-blind, placebo-controlled phase 1 trial. Hum Vaccin Immunother. 2022 Nov 30;18(6):2092363. doi: 10.1080/21645515.2022.2092363. Epub 2022 Jul 14. PMID 35834812